CLINICAL TRIAL: NCT00150358
Title: Open Label, Multicenter, Non Comparative Study, To Confirm The Efficacy And Tolerability Of Viagra In Subjects With Erectile Dysfunction And Arterial Hypertension Who Are Taking Antihypertensive Treatment.
Brief Title: To Yield Further Information On The Efficacy And Safety Of Viagra Among Subjects With Arterial Hypertension .
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481187
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence; Hypertension
MeSH Terms: conditions — Erectile Dysfunction; Hypertension | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate

SUMMARY:
To assess changes with respect to Erectile Dysfunction in subjects treated with Viagra and antihypertensive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with arterial hypertension treated with one or more antihypertensive agents, the doses of which have been stable for at least 4 weeks prior to the baseline visit, with a documented clinical diagnosis of ED and a confirmation of this by a qualification of 21 or less on the SHI-M.

Exclusion Criteria:

* Subjects with resting sitting systolic blood pressure >170 or <110mmHg or resting sitting diastolic blood pressure >90 or <50mmHg, with significant cardiovascular disease and retinitis pigmentosa, treatment with nitrates, alfablockers or CYP3A4 inhibitors.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253
Dates: Start 2005-03; Study Completion 2005-11

PRIMARY OUTCOMES:
The primary efficacy measure is the percent of ITT subjects at week 8 with positive response to the Global Efficacy Assessment question regarding the effectiveness of the medication in improving erections over no treatment at all for ED.

SECONDARY OUTCOMES:
The evaluation of change from baseline to week 8 on the toal SHI-M (Sexual Health Inventory-Male) score and the 5 individual items on the SHI-M. Global Efficacy Assessment Questions 2 and 3 at week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Mexico (15):
  - Pfizer Investigational Site, Torreón, Coahuila
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Colonia Centro, Mexico City
  - Pfizer Investigational Site, DF, Mexico City
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, San Luis PotosÃ-, San Luis PotosÃ-
  - Pfizer Investigational Site, Mérida, Yucatán
  - Pfizer Investigational Site, Aguascalientes
  - Pfizer Investigational Site, Chihuahua City
  - Pfizer Investigational Site, Durango
  - Pfizer Investigational Site, Metepec
  - Pfizer Investigational Site, Puebla City
  - Pfizer Investigational Site, San Luis Potosí City
  - Pfizer Investigational Site, Veracruz